CLINICAL TRIAL: NCT01822249
Title: A Phase 2A Randomized, Placebo Controlled Trial of EPI-743 in Children With Rett Syndrome
Brief Title: Phase 2 Study of EPI-743 for Treatment of Rett Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPBGC&RS_12_003
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; EPI-743; Edison
MeSH Terms: conditions — Rett Syndrome | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPI-743 15 mg/kg (Active Comparator): Subjects in this arm will receive EPI-743 at a dose of 15 mg/kg three times daily
  Interventions: Drug: EPI-743
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo at a volume equivalent to the volume of EPI-743 they would receive if in active group based on their weight
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EPI-743
  Arms: EPI-743 15 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Rett syndrome is a severe neurodevelopmental disorder that primarily affects female children. Rett syndrome is characterized by significant elevation in blood markers of oxidative stress. EPI-743 is a novel therapeutic with demonstrated efficacy and safety in the treatment of disorders characterized by oxidative stress. The purpose of this study is to examine the safety and efficacy of EPI-743 in a population of children with Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rett syndrome with disease stage 1-2
* Abnormality of at least two disease biomarker levels
* Confirmed MeCP2 mutation
* Patient or patient's guardian able to consent and comply with protocol requirements
* Abstention from use of Coenzyme Q10, vitamin E and Idebenone two weeks prior to enrollment into the study

Exclusion Criteria:

* Any condition, which in the opinion of the investigator could compromise the subject's safety or adherence to treatment with EPI-743.
* Clinically significant allergy or hypersensitivity to EPI-743 or to any of the excipients of with EPI-743 (eg., sesame oil).
* Clinically significant allergy or hypersensitivity to Vitamin E
* Lack of confirmation of MeCP2 mutation
* Clinical history of bleeding or abnormal baseline PT/PTT
* Diagnosis of any other concurrent inborn error of metabolism
* Hepatic insufficiency with LFTs greater than 3 times upper limit of normal
* Renal insufficiency requiring dialysis
* End stage cardiac failure
* Fat malabsorption syndromes precluding drug absorption

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Rett Syndrome Clinical Severity Sore | Change at six months from baseline
  Measure of disease progression

SECONDARY OUTCOMES:
Oxidative Stress Biomarkers | Change at six months from baseline
Head circumference | Change at six months from baseline
Rett syndrome behavioral questionnaire | Change at six months from baseline
PedsQL | Change at six months from baseline
Number of Drug-related adverse and serious adverse events | Six months
Respiratory Disturbance Index (RDI) | Change at six months from baseline
  RDI will be determined on polysomnography study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: No